CLINICAL TRIAL: NCT06593223
Title: Non-invasive Filling Pressure(NIFP) Device Based on Low Frequency Heart Sound in Assessment of Congestion in Heart Failure Patients
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Collaborators: Shenzhen Fiber Medical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 伦[2019]165
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute heart failure (AHF) patients: For acute heart failure (AHF) patients：NIFP test were conducted 2-3 times during the hospital stay. The first test is supposed to be conducted close to the time of admission. In the same day of each NIFP test a physical examination is performed to the patient and clinical congestion score (CCS) is recorded. If available, the Nt-proBNP test result in the same day of NIFP test is recorded. Echocardiography examination is scheduled for most of patients and Ejection Fraction (EF), E/A, and E/e' ratio are recorded as well.
  Interventions: Device: Assess Non-invasive filling pressure(NIFP) in heart failure patients
- Stabilized outpatient chronic heart failure patients: For stabilized outpatient chronic heart failure patients：NIFP test was conducted and if Nt-proBNP test result is available in the same day it will be recorded as well.
  Interventions: Device: Assess Non-invasive filling pressure(NIFP) in heart failure patients

INTERVENTIONS:
Device: Assess Non-invasive filling pressure(NIFP) in heart failure patients — Assess Non-invasive filling pressure(NIFP) in outpatients with stable heart failure and inpatients with acute heart failure in ward

SUMMARY:
Congestion plays a key role in heart failure (HF) trajectory .Clinical congestion refers to the signs and symptoms resulting from elevated cardiac filling pressures. Hemodynamic congestion refers to elevated cardiac filling pressures, which may occur days or weeks before the presentation of symptoms , , .

Serial assessment of congestion is required in each encounter of the HF patients, while in current clinical practice, serial assessment of congestion relies on physical examination, sometimes supported by BNP test. Both physical and BNP test are reported to be unreliable in some cases ， . Echocardiography is good tool, but it requires skilled physician to operation and is more time consuming. In general, there is unmet needs of better tools for serial assessment of congestion in HF patient management.

In this study, we aim to prospectively observe and evaluate the feasibility of using a novel non-invasive device in assessment of congestion in HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute heart failure；Stabilized outpatient chronic heart failure patients；Willing to sign the inform consent

Exclusion Criteria:

* 1.Patients under 18 years old 2.Patients with congenital heart diseases (e.g., tetralogy of Fallot, atrial septal defect, Fontan disease, single chamber disease) 3.Patients with implanted artificial mechanical valves, pacemaker or ICD. 4.Patients with significant back issues that prevent them from lying supine on the bed 5.Pregnant patients 6.Patient wight under 35 kg or over 150 kg 7.Patients who are attaching to other medical device that prevent them to receive a test by the study device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient visits to hospital with suspected heart failure (HF) or with history of HF were enrolled. Some of the patients were admitted to cardiology ward due to initial diagnosis of acute heart failure (AHF). Some of the patients are who make a planned visit to outpatient clinic with history of HF. All patients are over 18 years old and are willing to sign the inform consent.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Noninvasive filling pressure testing has clinical significance consistent with NT-proBNP and CCS scores to reflect congestion in acute heart failure. | 2025-7-1
  Noninvasive filling pressure testing has clinical significance consistent with NT-proBNP and CCS scores to reflect congestion in acute heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Mingya Liu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No